CLINICAL TRIAL: NCT02411097
Title: Prevention of Deep Venous Thromboembolism: Effect of Preemptive Analgesic of Femoral Nerve Block in Patients Undergoing Total Knee Arthroplasty
Brief Title: Role of Femoral Nerve Block on Prevention of Postoperative Deep Venous Thromboembolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CJGG2014
Record Dates: First submitted 2015-03-20; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-03

CONDITIONS: Gonarthrosis
Keywords: Deep venous thromboembolism; Femoral nerve block; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- femoral nerve block (Experimental): femoral nerve block will be administered before or after the surgery
  Interventions: Procedure: femoral nerve block

INTERVENTIONS:
Procedure: femoral nerve block — use the nerve stimulator,the femoral nerve block will be administered before or after the surgery

SUMMARY:
To investigate whether preemptive analgesic of femoral nerve block could prevent deep venous thromboembolism due to inhibiting the excessive release of neutrophil elastase and inflammatory cytokines.

DETAILED DESCRIPTION:
Femoral nerve block is an effective analgesic mode in patients after total knee arthroplasty. In recent studies, there has been shown that a large amount of neutrophil elastase release from neutrophils could induce the development of deep venous thromboembolism and femoral nerve block may reduce the incidence of the development of deep venous thromboembolism. In addition, inflammatory cytokines including interleukin-1(IL-1), IL-6, IL-8 and tumor necrosis factor(TNF) were associated with deep venous thromboembolism. Thus, the investigators hypothesised that preemptive analgesic of femoral nerve block could prevent deep venous thromboembolism due to inhibiting the excessive release of neutrophil elastase and inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for total knee arthroplasty under general anesthesia

Exclusion Criteria:

* ASA physical status Ⅳ-Ⅴ,
* psychiatric illness,
* chronic opioid consumption,
* patient refusal,
* coagulopathy,
* peripheral neurological injury,
* local anesthesia drug allergy,
* preoperative existing deep venous thromboembolism.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of inflammatory cytokine | change from baseline at 30min, 60min, 90min after using tourniquet and 12h, 24h,48h after operation

SECONDARY OUTCOMES:
Concentration of related inflammatory factors of deep venous thromboembolism | change from baseline at 30min, 60min, 90min after using tourniquet and 12h, 24h,48h after operation
  inflammatory factors include IL-1, IL-6, IL-8 and TNF，detecting the concentrations by enzyme-linked immunosorbent assay (ELISA).

OTHER OUTCOMES:
Diagnosis of deep venous thromboembolism by ultrasonography | 2day and 7day after operation
  result of diagnosis is yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wang, Principal Investigator — Gereral Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China